CLINICAL TRIAL: NCT03876951
Title: Prospective Multicenter Pilot Study to Evaluate the Accuracy of Percutaneous Biopsy by Vacuum-assisted Biopsy (VAB) to Assess Pathological Complete Response in Patients With Clinical and Radiological Complete Response After Neoadjuvant Chemotherapy (NeoVAB)
Brief Title: Evaluation of the Accuracy of Percutaneous Biopsy by Vacuum-assisted Biopsy (VAB) to Assess Pathological Complete Response in Patients With Clinical and Radiological Complete Response After Neoadjuvant Chemotherapy (NeoVAB)
Acronym: NeoVAB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NeoVAB
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Vacuum-assisted Biopsy
Keywords: breast cancer; neoadjuvant chemotherapy; vacuum-assisted biopsy; pathological complete response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vacuum-assisted biopsy (Experimental): Patients will be submitted to percutaneous vacuum-assisted biopsy (VAB), followed by breast surgery
  Interventions: Diagnostic Test: Vacuum-assisted biopsy

INTERVENTIONS:
Diagnostic Test: Vacuum-assisted biopsy — Patients will be submitted to percutaneous vacuum-assisted biopsy (VAB), followed by breast surgery.

SUMMARY:
Breast cancer is the most commonly diagnosed cancer and the leading cause of cancer death in females in the world. Neoadjuvant chemotherapy (NAC) is increasingly used in patients with operable breast cancer to enhance the likelihood of breast conservation. New generation of treatments or combinations lead to a high rate of pathological complete responses (pCR) in patients with human epidermal growth factor receptor 2 positive (HER2) and triple negative tumours. Safe omission of surgery in patients who receive NAC and achieve radiologic complete response depends on the ability to accurately estimate pCR preoperatively.

If pathological complete response after NAC could be accurately assessed by VAB, surgery could be avoided. In the context of new treatments or combinations with an increased pCR rate, this new strategy could induce major changes in clinical practice, leading to breast surgery de-escalation.

DETAILED DESCRIPTION:
A total of 66 patients will be submitted to percutaneous vacuum-assisted biopsy (VAB), followed by breast surgery. The primary endpoint of the study is the false negative rate of VAB procedure. This rate will be calculated by comparing the detection of invasive or in situ carcinoma on surgical specimen versus VAB samples. The secondary endpoints of the study are feasibility, VAB procedure technical complications and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older.
2. Written informed consent provided.
3. Triple negative or HER2-positive / ER-negative or HER2-positive / ER-positive breast tumours.
4. Patients eligible for breast conservation after NAC.
5. Patients with T2-T3 N0 invasive breast cancer initially treated by NAC to allow breast conservation, who have received a minimum of 6 cycles of adequate NAC +/- anti-HER2.
6. Clinical complete response after NAC.
7. Radiological (mammography, breast US, breast MRI) complete response after NAC.
8. Patients predicted to be node-negative at treatment initiation.

Exclusion Criteria:

1. Patient younger than 18 years old.
2. Pregnant or breastfeeding women.
3. Proven metastatic axillary or internal mammary chain lymph node involvement before NAC proven by biopsy or cytology.
4. Bilateral breast cancer.
5. Contraindication to MRI.
6. Contraindication to breast conservation
7. Patients with a BRCA mutation or other autosomal dominant high-penetrance genetic predisposition to breast cancer.
8. Patients with limitation of freedom or under guardianship
9. Inability for psychological reasons
10. Hypersensitivity to local anaesthesia
11. Initial imaging showing ACR6 micro calcifications and/or ACR6 non-mass enhancement associated to the index lesion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
False negative rate of vacuum-assisted biopsy | During the surgery
  Absence of invasive and in-situ carcinoma on vacuum-assisted biopsy but presence of invasive or in-situ carcinoma on the surgical specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France